CLINICAL TRIAL: NCT07399587
Title: Optimizing the Management of Patients With Heart Failure With Reduced Ejection Fraction Using BaroStim and CardioMems
Brief Title: Optimizing HFrEF Patients Using BaroStim and CardioMems
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0583
Record Dates: First submitted 2025-12-22; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure NYHA Class III
Keywords: NYHA Class III heart failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BaroStim (Experimental): The intervention is insertion and titration of BaroStim. This is for patients with NYHA Class III heart failure who are candidates for CardioMems insertion (or have already received CardioMems in the past 3 months) and subsequent BaroStim insertion.
  Interventions: Device: BaroStim

INTERVENTIONS:
Device: BaroStim — BaroStim NEO or BaroStim NEO2 will be used in this study. The device consists of a Carotid sinus lead 2 mm in thickness and an implantable pulse generator. The study intervention is monitoring of CardioMems reading while titrating the BaroStim device.

SUMMARY:
The goal of this study is to utilize CardioMems (measurement of pulmonary artery diastolic pressure) to assess BaroStim. At the time of CardioMems insertion, patients will be screened for candidacy to receive a BaroStim device. Patients will be followed for 3 months after the CardioMems insertion before undergoing insertion of a Barostim. Patients who have undergone a CardioMems, will be eligible for enrollment after 3 months of medication management and optimization. Patients will be followed for 1 year after insertion of Barostim.

DETAILED DESCRIPTION:
This is a longitudinal, single arm study in which patients will serve as their own controls prior to study intervention (BaroStim insertion). All patients eligible for both CardioMems and BaroStim devices will undergo insertion per standard of care, regardless of participation in this study. After placement of CardioMems, patients will undergo 3 months of medication management and titration. After 3 months of medication titration, patients will undergo BaroStim insertion. This sequential placement of devices along with the 3 month medication titration period is standard of care and will occur prior to enrollment in the study. Subsequently, patients will be seen for in-office visits for titration of BaroStim along with measurement of pulmonary artery diastolic pressure, 6MWT, and vital signs. The goal will be to achieve a pulmonary artery diastolic pressure (PADP) of 18-20 mm Hg or less. Patients will be followed for up to 1-year post-insertion.

The goal of this study is to utilize the pulmonary artery diastolic pressure (obtained from CardioMems) as an objective method to assess BAT. A 10% improvement in 6MWT, blood pressure, PADP, NT pro-BNP, or LVEF, or any improvement in NYHA class is deemed clinically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ages 18-80 years
4. Diagnosed with NYHA Class III Heart Failure with LVEF<35%
5. Able to tolerate oral medications for guideline directed medical therapy titration period
6. Have undergone insertion of CardioMems and BaroStim devices per standard of care.
7. It is a standard of care to recommend that females of reproductive potential use highly effective contraception, because of the teratogenic potential of many medications used to treat HFrEF. In addition, withdrawal of GDMT during pregnancy may reverse the positive remodeling and lead to life threatening worsening of heart failure. Women of child-bearing age need to agree to use such a method during study participation and indefinitely after the end of the study.

Exclusion Criteria:

1. Individuals ineligible for either CardioMems or BaroStim devices.
2. NT-proBNP >1600 mg/dL
3. Indicated for CRT-D device (left bundle branch block)
4. Initial 6-minute walk test distance less than 140 m
5. Left ventricular assist device (LVAD)
6. History of carotid vascular procedure (carotid endarterectomy)
7. Pregnancy or lactation
8. Known allergic reactions to components of the BaroStim or CardioMems insertion or guideline directed medical therapy for heart failure
9. Febrile illness within 30 days of study enrollment
10. Treatment with another investigational drug or other intervention within 1 year
11. Current smoker or tobacco use within 1 year
12. Enrolled in any other CVRx funded study, including investigator-initiated research, registries, or other pre- or post-market studies.
13. Vulnerable individuals as outlined below

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Artery Diastolic Pressure | During procedure
  Pulmonary Artery Diastolic Pressure as Measured by CardioMems Device
6 Minute Walk Test | Through study completion, 1 year
  Distance covered in 6 minute walk test
Blood Pressure | Through study completion, 1 year
  Systolic and diastolic blood pressure at repeated clinic visits
NYHA Class of Heart Failure | Through study completion, 1 year
  Any change or improvement of NYHA Class of Heart Failure
NT-pro BNP Levels | Through study completion, 1 year
  Any change or improvement of NT-pro BNP levels
LVEF | Through study completion, 1 year
  Any change or improvement in LVEF
Medication Usage | Through study completion, 1 year
  Any change or improvement in medication usage

SECONDARY OUTCOMES:
Incidence of Hospitalizations | Through study completion, 1 year
  Incidence of hospitalizations for acute decompensated heart failure during study period.

CONTACTS AND LOCATIONS:
Overall Officials: John Kassotis, MD, Principal Investigator — Northwell Health
Locations (1):
- Peconic Bay Medical Center, Riverhead, New York, United States